CLINICAL TRIAL: NCT05273138
Title: Analysis of Dermal Fibroblasts and Immune Cells During Systemic Sclerosis
Acronym: Skin-SSC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0611; 2021-A03137-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Fibrosis, fibroblasts.; Fibroblasts.; Immune system.; B lymphocytes.
MeSH Terms: conditions — Scleroderma, Systemic; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic sclerosis patients: Patients fulfilling the ACR/EULAR criteria for systemic sclerosis
  Interventions: Other: Blood sampling and skin biopsy
- Healthy subjects
  Interventions: Other: Blood sampling and skin biopsy

INTERVENTIONS:
Other: Blood sampling and skin biopsy — Blood sampling and skin biopsy

SUMMARY:
The pathophysiology of systemic sclerosis (SSc) is still poorly understood and there are no effective treatments for this disease. SSc is a heterogeneous disease with varying severity. The heterogeneity of fibroblast profiles, observed in other fibrosing pathologies, has never been thoroughly explored in the skin of SSc patients. The immune system, and in particular B lymphocytes, plays a central role in the pathophysiology of SSc. The interactions between B lymphocytes and the cells responsible for excess collagen production, i.e. fibroblasts, are not fully elucidated The main objective is to analyze the heterogeneity of fibroblasts and infiltrating immune cells as well as their molecular signature in the skin of patients with SSc

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years of age
* With a systemic sclerosis meeting the ACR-EULAR 2013 criteria Having signed an informed consent
* Being insured

Exclusion Criteria:

* Syndrome of overlap with another connective tissue disease according to the international diagnostic criteria
* Immunosuppressive treatment within 12 months
* Dosage of current corticosteroid therapy ≥10mg/d
* Protected minors or adults
* Pregnant or breastfeeding women
* Deprived of their liberty
* Persons in emergency situations
* Persons who have refused or are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the University Hospital of Lille
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Single cell RNAseq transcriptomic analysis of skin | At inclusion

SECONDARY OUTCOMES:
Single cell RNAseq transcriptomic analysis of the whole blood | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France